CLINICAL TRIAL: NCT00956280
Title: Epidemiologic Study of KRAS Mutation in Brazilian Patients With Advanced or Metastatic Non Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Laboratorio Progenetica (Unknown)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-OBR-DUM-2008/1; IMPACT 14829
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2010-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: The frequency and type of KRAS mutation in a sample of the Brazilian population with advanced NSCLC; KRAS mutation in population with advanced NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to characterize the demographic and clinical aspects, and describe the frequency and type of KRAS mutation in a Brazilian population sample with advanced non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of locally advanced or metastatic Non Small Cell Lung Cancer (IIIB-IV)
* Tumour sample (block of slides) available for KRAS analysis

Exclusion Criteria:

* Confirmation of locally advanced or metastatic NSCLC (IIIB-IV) exclusively by cytology, with no tumour sample access.
* Previous treatment using a MEK inhibitor or any other regimen containing docetaxel (previous treatment with paclitaxel is accepted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Advanced Non Small Cell Lung Cancer
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To analyze the frequency and type of KRAS mutation in a sample of the Brazilian population with advanced NSCLC. | March 31, 2010

CONTACTS AND LOCATIONS:
Overall Officials: José Eduardo Pipolo das Neves, MD, Study Director — AstraZeneca do Brasil, MC Medical Director
Locations (5):
- Brazil (5):
  - Research Site, Belo Horizonte
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santo André
  - Research Site, São Paulo